CLINICAL TRIAL: NCT01460004
Title: The Effect of Infra Patellar Strap Treatment on the Extent of Pain and Performance in Young Athletes With Patellar Tendinopathy
Brief Title: The Effect of Infrapatellar Strap Treatment on Pain Extent and Athletic Measures in Young Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wingate Institute (Other)
Responsible Party: Principal Investigator, Dr. Eyal Shargal, Professional director, Sports Medicine Sciences and Research,, Wingate Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Winphys01
Record Dates: First submitted 2011-10-05; First posted 2011-10-26 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Patellar Tendonitis; Jumper's Knee; Patellar Tendinopathy
Keywords: patellar tendinopathy; jumper's knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patella knee strap (No Intervention): infra patella knee strap- cotton, applied in straight leg
  Interventions: Device: patella knee strap

INTERVENTIONS:
Device: patella knee strap — infra patella strap 100% cotton pressure is exerted immediately under the patella
  Other Names: FDA regulation number 890.3475

SUMMARY:
The purpose of this study is:

* To examine the effect of infra patellar strap treatment on the extent of pain and jumping performance tasks in young male athletes diagnosed with patellar tendinopathy.
* 40 elite male athletes, basketball and volleyball players, ages 14-18, students of the academy for sports Excellency will take part in this study
* Hypothesis 1: The treatment of infra patellar strap will reduce the level of pain during jumping performance tasks.
* Hypothesis 2: The treatment of infra patellar strap will improve the squat jump height in athletes with patellar tendinopathy during squat jump task.
* Hypothesis 3: The treatment of infra patellar strap will improve the drop jump height in athletes with patellar tendinopathy during drop jump task.
* Hypothesis 4: The treatment of infra patellar strap will improve the one leg jump height in athletes with patellar tendinopathy during one leg jump task.
* Hypothesis 5: The treatment of infra patellar strap will improve the 30 seconds repetitive jumps mean height in athletes with patellar tendinopathy during 30 seconds repetitive jumps task.

DETAILED DESCRIPTION:
Introduction: Patellar tendinopathy (Jumper's knee) is a condition usually characterized by localized pain and tenderness of the patellar tendon at its origin on the inferior pole of the patella.

Patellar tendinopathy is an over use injury which implies on a mismatch between stress on a given tissue and the ability of that tissue to withstand the stress. Rapid repetitive actions of acceleration, deceleration, jumping and landing place great stress on the extensor mechanism and the patellar tendon.

Current prevalence reported of patellar tendinopathy is up to 20% among elite athletes from a range of sports, with higher proportions in professional basketball (32%) and volleyball (45%) players.

The common treatment for patellar tendinopathy is preventative or conservative (physical therapy).

Infra patellar straps are used in treatment to reduce anterior knee pain from a variety of sources including patellar tendinopathy, patellar subluxation, patellar femoral syndrome, Osgood-Schlatter disease and more.

In spite of the frequent use of this strap in young athletes and the subjective report of decreased anterior knee pain experienced by the athletes using them, the mechanisms for reducing anterior knee pain has not been explained.

In addition, there is no data on the straps effect regarding the extent of pain and functional performance as jumping in this population.

The purpose of this study: To examine the effect of infra patellar strap treatment on the extent of pain and jumping performance tasks in young male athletes diagnosed with patellar tendinopathy.

Methods: 20 elite male athletes, basketball and volleyball players, ages 14-18, students of the academy for sports Excellency will take part in this study. Athletes approaching the physical therapy department of the Ribstein Center for Sport Medicine Sciences and Research at Wingate Institute, with anterior knee pain, will be examined by a professional physical therapist. The ones who are diagnosed with chronic patellar tendinopathy will be included in the study.

Each athlete will attend one meeting in which he will perform four tests: Squat jump test, Drop jump test, one leg jump test and jumps 30 seconds test. The tests with and without the infra patellar strap will be performed using The Optojump measuring system (Microgate, Bolzano, Italy). In addition the athlete will grade his pain severity with and without the infra patellar strap, using The Visual Analog Scale (VAS).There will be no follow up, all the data will be collected in one session.

Data will be collected between january 2012 and december 2012, data analysis and summary of the study will be finished at december 2013.

Statistical Analysis: In order to examine the difference between the tests results with and without the infra patellar strap, dependent t- test will be performed. Significant level will be set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* elite male athlete
* basketball and volleyball player
* ages 14-18
* clinical diagnosis of patellar tendinopathy
* able to jump

Exclusion Criteria:

* undergo a surgical procedure in knee

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
change in pain level after applying an infra patellar strap | Within a week from primary physical therapist examination and including in the study. Measures will be taken Before, during and after jump tasks with and without the infra patelar strap, during one session.
  level of pain ranked upon visual analog scale by the subject

SECONDARY OUTCOMES:
change in height of jump after applying an infra patellar strap | Within a week from primary physical therapist examination and including in the study. while performing the jumps tasks with and without the infra patellar strap. All measures will be collected during one session, without follow-up.
  the height of squat jump, drop jump, one leg jump and 30 sec repetitve jumps (mean height) as mesured by the optojump system

CONTACTS AND LOCATIONS:
Overall Officials: gali dar, Phd, Study Director — Wingate Institute
Locations (1):
- Wingate Institute, Netanya, Israel